CLINICAL TRIAL: NCT01445028
Title: Determining the Effect of Low-dose Isotretinoin on Proliferative Vitreoretinopathy
Brief Title: Isotretinoin for Proliferative Vitreoretinopathy
Acronym: DELIVER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Richard S. Kaiser, Associate Clinical Professor, Wills Eye
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WEI-DELIVER
Record Dates: First submitted 2011-09-29; First posted 2011-10-03 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-04

CONDITIONS: Proliferative Vitreoretinopathy
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Isotretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Primary, high-risk retinal detachment (Experimental): Oral isotretinoin on recurrent retinal detachment associated with Proliferative vitreoretinopathy
  Interventions: Drug: Isotretinoin
- Recurrent RD associated with PVR (Experimental): Oral isotretinoin on recurrent retinal detachment associated with Proliferative vitreoretinopathy
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin 20mg daily for 12 weeks

SUMMARY:
Proliferative vitreoretinopathy (PVR), or secondary scarring on and around the retina, is an important cause of retinal re-detachment. The purpose of this study is to evaluate the effect of oral isotretinoin, which inhibits the growth of cells responsible for proliferative vitreoretinopathy (PVR), on recurrent retinal detachment.

DETAILED DESCRIPTION:
Small retrospective studies have shown isotretinoin to be effective in reducing the rate of recurrent retinal detachment in patients with or at high risk for developing PVR. This is a prospective study to evaluate a low dose of oral isotretinoin in this regard. There are two arms to the study: 1) eyes with recurrent retinal detachment due to existing PVR, and 2) eyes with primary detachment and features associated with a high risk of PVR formation. Eligible and willing patients will receive a 12-week course of isotretinoin, and will be followed for retinal attachment rate, and PVR and/or ERM (epiretinal membrane) formation.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 year-old men or 50-70 year-old, post-menopausal women.
* Healthy enough to participate in the study.
* Willing and able to consent to participation.
* Recurrent PVR-associated RD occurring at least 2 weeks after RD repair or
* Primary RD (retinal detachment) associated with one or more high-risk features

Exclusion Criteria:

* History of hypersensitivity to isotretinoin.
* Current use of a corticosteroid (excluding topical).
* Any history of depression, anorexia, liver or pancreatic disease.
* More than one prior surgical RD repair.
* Patients with closed funnel retinal detachments.
* Patients with chronic retinal detachment, defined as longer than 12 weeks.
* Any use an oral retinoid within 6 months.
* Systemic chemotherapy within 6 months.
* Patients taking supplemental vitamin A.
* Corneal opacity sufficient to impair surgical view.
* Proliferative diabetic retinopathy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2011-09; Primary Completion 2013-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Kaiser, MD, Principal Investigator — Wills Eye Institute
Locations (1):
- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary, High-risk Retinal Detachment | Recurrent RD Associated With PVR
Started | 58 | 54
Completed | 58 | 51
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary, High-risk Retinal Detachment | Recurrent RD Associated With PVR | Total
Number analyzed (Participants) | 58 | 51 | 109
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 51 | 35 | 86
  >=65 years | 7 | 16 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (10.0) | 59.7 (11.8) | 57.1 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 11 | 26
  Male | 43 | 40 | 83
Region of Enrollment [Number; unit: participants]
  United States | 58 | 51 | 109

OUTCOME MEASURES:

1. Primary Outcome: Rate of Retinal Attachment
Description: We will evaluate all patients for retinal attachment at 3 months.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Primary, High-risk Retinal Detachment | Recurrent RD Associated With PVR
Number analyzed (Participants) | 58 | 51
Participants | 50 | 42

ADVERSE EVENTS:
Arm/Group | Primary, High-risk Retinal Detachment | Recurrent RD Associated With PVR
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/54
Other Adverse Events (participants affected / at risk) | 0/58 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes